CLINICAL TRIAL: NCT05256849
Title: Treatment of Humeral Fractures With Long PHILOS Plates Using a Modified Technique and Approach Avoids Radial Nerve Palsy
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-01959; mu22Rikli
Record Dates: First submitted 2022-02-16; First posted 2022-02-25 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Humeral Fracture
Keywords: PHILOS plate; minimal invasive plate osteosynthesis (MIPO); radial paralysis
MeSH Terms: conditions — Humeral Fractures; Paralysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Radial paralysis is a well-known complication of plate osteosynthesis on the humeral shaft. At the University Hospital Basel, these fractures have been treated in an adapted procedure with long PHILOS plates using a modified technique and approach. This study is to retrospectively analyze the effectiveness of the surgical technique in relation to iatrogenic radial paralysis.

DETAILED DESCRIPTION:
Radial paralysis is a well-known complication of plate osteosynthesis on the humeral shaft. With regard to surgical treatment, there are major differences in terms of surgical access and implant selection. At the University Hospital Basel, these fractures have been treated in an adapted procedure for about 10 years. A long Philosplatte (Synthes company) is inserted from the proximal end via a deltoido-pectoral approach. This is a minimally invasive procedure (MIPO = minimally invasive plate osteosynthesis). The standard implant is first twisted distally by approx. 45°-90° and then lies anterior to the humerus. The distal screws can then be filled via anterior stab incisions. This adapted surgical technique is adapted to the anatomical course of the radial nerve. This ensures a safe distance from the plate/access to the nerve. The nerve does not have to be explored openly and the distal row of screws can be used minimally invasively via stab incisions. This study is to retrospectively analyze the effectiveness of the surgical technique in relation to iatrogenic radial paralysis.

ELIGIBILITY:
Inclusion Criteria:

* surgery at the University Hospital Basel between 06/2010 and 12/2020 for a proximal humeral shaft fracture

Exclusion Criteria:

* Patients with a documented rejection

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients aged 18 and over who underwent surgery at the University Hospital Basel between 06/2010 and 12/2020 for a proximal humeral shaft fracture
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
descriptive statistical analysis of datasets from patients treated with the adapted surgical technique | one time assessment at baseline
  datasets from patients (information about hospitalizations and risk factors, traumatological and orthopedic information (precise diagnosis and classification, date, number and type of operation, complications), infectious data (detection of germs, type and duration of therapy)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Rikli, Prof. Dr. med., Principal Investigator — University Hospital Basel, Clinic for Orthopedics and Traumatology
Locations (1):
- University Hospital Basel, Orthopedics and Traumatology, Basel, Switzerland